CLINICAL TRIAL: NCT01940302
Title: Metabolic Control Before and After Supplementation With LEHEL in Patients With Type 2 Diabetes
Brief Title: Dietary Supplement of LEHEL for the Patients With Type 2 Diabetes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shaoguan University (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGU-03; 2012BAD33B10 (Other: National Key Technology Research and Development Program of China)
Record Dates: First submitted 2013-09-07; First posted 2013-09-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Type 2 Diabetes
Keywords: Malnutrition; Metabolic disorders
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Malnutrition; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LEHEL multi-nutrients supplement (Experimental): 75 g/d of LEHEL supplementation along with oral hypoglycemic agents such as glibenclamide and/or metformin.
  Interventions: Dietary Supplement: LEHEL multi-nutrients supplement
- Control (No Intervention): Received only oral hypoglycemic agents.

INTERVENTIONS:
Dietary Supplement: LEHEL multi-nutrients supplement — The primary objective of this study is to evaluate the effect of a diet program including LEHEL multi-nutrients supplement as breakfast replacement on metabolic control after 12-week intervention in subjects with type 2 diabetes.
  Arms: LEHEL multi-nutrients supplement

SUMMARY:
Due to metabolic disorders and dietary restrictions, patients with diabetes may have different degrees of malnutrition. The primary objective of this study is to investigate whether supplementation of LEHEL, a multi-nutrients supplement, is capable to improve metabolic parameters in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with type 2 diabetes mellitus according to the Chinese type 2 diabetes prevention guide 2010, diagnostic criteria are as follows:

  (1) Diabetes symptoms（polydipsia、polyphagia, polyuria, weight loss、skin itching、blurred vision and other acute metabolic network disorder that caused by high blood sugar）combined with random blood sugar ≥11.1 OR, (2) fasting plasma glucose (FPG) ≥7.0 OR, (3) 2 h blood sugar after oral glucose tolerance test (OGTT) ≥11.1;
* Subject is between 18 and 75 years of age, inclusive.
* Subject's BMI is >18.5 kg/m2 and <35 kg/m2.
* If on a chronic medication such as anti-hypertensive, lipid-lowering, thyroid medication or hormone therapy, subject has been on constant dosage for at least two months prior to screening visit.

Exclusion Criteria:

* Subject that is diagnosed as type 1 diabetes, gestational diabetes and other kinds of diabetes expect type 2.
* Subject that use exogenous insulin for glucose control.
* Subject that has a history of diabetic ketoacidosis.
* Subject that has mental disorder, cancer, cirrhosis, renal disease and hepatic disease.
* Subject that has had a significant cardiovascular event less than six months prior to screening visit or has history of congestive heart failure.
* Subject that has had operation less than six months prior to screening visit.
* Subject that has taken/is currently taking any dietary supplements or medications that could profoundly affect blood glucose during the past one month prior to screening visit.
* Subject is known to be allergic or intolerant to any ingredient found in the study product.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Metabolic Control | Twelve weeks
  Hemoglobin A1c (HbA1c) and lipids (Cholesterol, HDL-cholesterol, Triglycerides) at study entry and 12 weeks after dietary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Wenhua Ling, Ph.D., Study Director — Sun Yat-sen University
Locations (1):
- Shaoguan University, Shaoguan, Guangdong, China